CLINICAL TRIAL: NCT04856163
Title: The Impact of Telelactation Services on Breastfeeding Outcomes: Digital Tele-MILC Trial
Brief Title: The Impact of Telelactation Services on Breastfeeding Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01NR018837 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding
Keywords: telehealth; telemedicine; health equity; disparities; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telelactation support (Experimental): Participants in the experimental group will receive unlimited, free telelactation visits with lactation consultants (IBCLCs) as demanded up to 24 weeks post-partum. Services will be available through mobile phone app.
  Interventions: Behavioral: Telelactation support
- ebook (No Intervention): Participants in the control arm will receive care as usual. They will also receive a ebook with content on infant care.

INTERVENTIONS:
Behavioral: Telelactation support — Participants will get unlimited access (through 24 weeks postpartum) to video calls with lactation consultants who are available 24/7. Participants can use the service as demanded.
  Arms: Telelactation support

SUMMARY:
This project will assess the impact of a novel breastfeeding support intervention ("telelactation"), delivered via video calls on personal devices including mobile phones and tablets. The goal of this intervention is to increase access to International Board Certified Lactation Consultants to improve, and reduce disparities in, breastfeeding rates. By implementing a digital randomized controlled trial that recruits participants through a popular pregnancy tracker mobile phone application, this mixed methods study will recruit a national sample of 1800-2400 individuals (depending on rate of attrition) during their third trimester of pregnancy to 1) provide evidence on the effectiveness of a widely available, yet understudied, service and 2) leverage technology to promote one of the most widely recommended health behaviors to improve children's health and to reduce disparities in key maternal and child health outcomes.

DETAILED DESCRIPTION:
This study is a pragmatic, parallel design randomized controlled trial that will generate evidence on the impact of telelactation on breastfeeding duration and exclusivity and explore differences in effectiveness by race/ethnicity. The study is mixed methods, and uses a sequential explanatory design in which qualitative interviews are used to explain and contextualize findings from the quantitative outcomes analysis. We will recruit primiparous, pregnant individuals age > 18 who intend to breastfeed and live in states most underserved by IBCLCs. Recruitment will occur via Ovia, a pregnancy tracker mobile phone application (app) used by one million pregnant individuals in the U.S. annually. Participants will be randomized to: 1) on-demand telelactation video calls on personal devices or 2) ebook on infant care/usual care. Breastfeeding outcomes will be captured via surveys and interviews and compared across racial and ethnic groups. This study will track participants for eight months (including six months postpartum), generating 1) quantitative data on the impact of telelactation and differences in effectiveness across racial and ethnic minority groups; and 2) rich qualitative data on the experiences of different subgroups of parents with the intervention, including barriers to use, satisfaction, and strengths and limitations of this delivery model.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* pregnant with first child
* intend to attempt breastfeeding
* residing in a state underserved by IBCLCs

Exclusion Criteria:

* non-singleton pregnancy
* advised by healthcare provider not to breastfeed for a medical reason (e.g., HIV+ status, chemotherapy planned)
* in police custody or incarcerated
* infant to be separated from birthing parent (e.g., given up for adoption, military deployment)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2108 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RAND Corporation, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from the proposed research will be shared with external researchers who request access beginning one year after the project ends. Results will be available to other researchers, public health workers, healthcare professionals, and community leaders who are interested in exploring approaches to improving breastfeeding rates following a brief application process. Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH. External researchers interested in investigator data, survey instruments, and other research methodology and procedures will obtain this information through collaborative agreements (e.g., data use agreements) with the principal investigator and co-investigators, as required by NIH's data sharing policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2025-2028

REFERENCES:
- [Derived] Uscher-Pines L, Kapinos K, Waymouth M, Howell K, Alvarado G, Ray K, Demirci J, Mehrotra A, Rogers R, James KF, DeYoreo M. Telelactation Services and Breastfeeding by Race and Ethnicity: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2461958. doi: 10.1001/jamanetworkopen.2024.61958. PMID 40014345
- [Derived] Uscher-Pines L, Demirci J, Waymouth M, Lawrence R, Parks A, Mehrotra A, Ray K, DeYoreo M, Kapinos K. Impact of telelactation services on breastfeeding outcomes among Black and Latinx parents: protocol for the Tele-MILC randomized controlled trial. Trials. 2022 Jan 3;23(1):5. doi: 10.1186/s13063-021-05846-w. PMID 34980212

RESULTS

PARTICIPANT FLOW:
Groups:
- Telelactation Support: Participants in the experimental group received unlimited, free telelactation visits with lactation consultants (IBCLCs) as demanded up to 24 weeks post-partum. Services were available through mobile phone app.
- Ebook: Participants in the control arm received care as usual. They will received a ebook with content on infant care.
Period: Overall Study
Arm/Group | Telelactation Support | Ebook
Started | 1052 | 1056
Completed | 955 | 956
Not Completed | 97 | 100
Not completed — Lost to Follow-up | 97 | 100

BASELINE CHARACTERISTICS:
Groups:
- Ebook: Participants in the control arm received care as usual. They also received an ebook with content on infant care.
- Total: Total of all reporting groups
Arm/Group | Telelactation Support | Ebook | Total
Number analyzed (Participants) | 1052 | 1056 | 2108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1052 | 1056 | 2108
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1052 | 1056 | 2108
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 383 | 380 | 763
  Not Hispanic or Latino | 669 | 676 | 1345
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 23 | 58
  Asian | 49 | 48 | 97
  Native Hawaiian or Other Pacific Islander | 9 | 6 | 15
  Black or African American | 301 | 310 | 611
  White | 509 | 474 | 983
  More than one race | 149 | 195 | 344
  Unknown or Not Reported | 0 | 0 | 0
Health insurance [Count of Participants; unit: Participants]
  Medicaid or Uninsured | 323 | 312 | 635
  Commercial or Other | 729 | 744 | 1473

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding Duration 1
Description: Number of participants who report any breastfeeding at 6 months
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Telelactation Support: Participants in the experimental group received unlimited, free telelactation visits with lactation consultants (IBCLCs) as demanded up to 24 weeks post-partum. Services were be available through mobile phone app.
- Ebook: Participants in the control arm received care as usual. They also received a ebook with content on infant care.
Arm/Group | Telelactation Support | Ebook
Number analyzed (Participants) | 955 | 956
Participants | 674 | 639
Statistical Analysis 1: Comparison: Telelactation Support vs Ebook; Test type: Superiority; p = 0.08, Regression, Logistic

2. Primary Outcome: Breastfeeding Duration 2
Description: Time to cessation of breastfeeding in months (as measured by reported age of infant when completely stopped receiving breastmilk)
Time Frame: 6 months post-partum
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Telelactation Support | Ebook
Number analyzed (Participants) | 955 | 956
months | 4.4 (2) | 4.5 (2)
Statistical Analysis 1: Comparison: Telelactation Support vs Ebook; Test type: Superiority; p = 0.21, discrete-time survival model

3. Primary Outcome: Breastfeeding Exclusivity
Description: Number of participants who report no formula use at 6 months
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Telelactation Support | Ebook
Number analyzed (Participants) | 955 | 956
Participants | 448 | 422
Statistical Analysis 1: Comparison: Telelactation Support vs Ebook; Test type: Superiority; p = 0.28, Regression, Logistic

4. Secondary Outcome: Breastfeeding Satisfaction
Description: Breastfeeding satisfaction at 6 months postpartum. Score on five-item maternal/infant breastfeeding satisfaction scale (which is a subscale of the Hill and Humenick lactation scale). Higher values indicate more agreement with the measures of satisfaction, resulting in a composite satisfaction score ranging from 5 to 25 for the subscale.
Time Frame: 6 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telelactation Support | Ebook
Number analyzed (Participants) | 952 | 956
score on a scale | 19.49 (5.43) | 18.95 (5.60)
Statistical Analysis 1: Comparison: Telelactation Support vs Ebook; Test type: Superiority; p = 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Telelactation Support | Ebook
All-Cause Mortality (participants affected / at risk) | 0/1052 | 0/1056
Serious Adverse Events (participants affected / at risk) | 0/1052 | 0/1056
Other Adverse Events (participants affected / at risk) | 0/1052 | 0/1056

LIMITATIONS AND CAVEATS:
Generalizability: Digital trials may not reach individuals without reliable access to technology and digital literacy; Inclusion criteria: We were not able to assess the impact of telelactation on breastfeeding initiation because we only enrolled individuals who intended to breastfeed; Outcomes were self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT04856163/Prot_SAP_000.pdf